CLINICAL TRIAL: NCT06775964
Title: Mesenchymal Stem Cell Therapy for Early Alzheimer's Disease
Brief Title: Stem Cell Therapy for Early Alzheimer's Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Paul E Schulz (Other)
Collaborators: Weston Brain Institute (Other)
Responsible Party: Sponsor-Investigator, Paul E Schulz, Principal Investigator, Director, Memory Disorders and Dementia Clinic, Professor of Neurology, Professor of Neurodegenerative Disorders, The University of Texas Health Science Center, Houston
Organization: The University of Texas Health Science Center, Houston (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-24-0516
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cognitive Dysfunction
Keywords: Mild Cognitive Impairment; Cognitive Decline; Alzheimer's disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: This is a Phase 1b/2a open label study to assess the safety and tolerability, as well as reduction of neuroinflammation after four IV-infusions of autologous, adipose-derived, Mesenchymal Stem Cells (adMSCs) over a 13-week treatment period in 12 subjects who are clinically diagnosed with late pre-symptomatic or prodromal AD, exhibit an Alzheimer's pathology and peripheral inflammatory profile.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- adMSC (Experimental): IV-infusions of autologous, adipose-derived, Mesenchymal Stem Cells (adMSCs)
  Interventions: Biological: adMSC

INTERVENTIONS:
Biological: adMSC — IV-infusion of autologous, adipose-derived, Mesenchymal Stem Cells (adMSCs), of approximately 2x10(8) adMSCs in 250mL saline.

SUMMARY:
The goal of this clinical trial is to learn if stem cell therapy works to treat brain inflammation in adults. Inflammation in the brain may be involved in adults who have memory or thinking problems. The stem cells will be taken from participant's fat samples, processed and given back to participants, so they are their own donor. The main questions this trial aims to answer are:

* Does stem cell therapy reduce inflammation in the brain?
* Does stem cell therapy improve brain activity?
* Does stem cell therapy slow down progression to Alzheimer's disease?

Participants will:

* Have a small fat biopsy taken at a doctor's office to process stem cells
* Receive 4 infusions of stem cells, through a vein in the arm over 12 weeks
* Visit the clinic every 2-4 weeks for the first 4 months and then every 1-2 months for 8 months for checkups and tests

DETAILED DESCRIPTION:
This is a Phase 1b/2a open label study to assess the safety and tolerability, as well as reduction of neuroinflammation after four IV-infusions of autologous, adipose-derived, Mesenchymal Stem Cells (adMSCs) over a 13-week treatment period in 12 subjects who are clinically diagnosed with late pre-symptomatic or prodromal AD, exhibit an Alzheimer's pathology and peripheral inflammatory profile.

To date, most drugs for AD primarily treat symptoms. Moreover, several anti-amyloid antibodies have reduced amyloid burden, but have only modestly affected cognitive progression, suggesting that other pathways are also important for AD progression. Neuroinflammation may be important for AD progression. The discovery of increased levels of inflammatory markers in patients at different clinical stages of AD, and the iden-tification of AD risk genes associated with innate immune functions, suggest that neuroinflammation may affect AD pathogenesis, making it an optimal candidate for targeted therapy to reduce disease progression. In this study, we aim to treat neuroinflammation with autologous adMSCs. These cells may represent a superior therapeutic alternative for AD be-cause they exhibit multi-therapeutic effects, including anti-inflammatory properties, reduced amyloid-β activity, and neurogenesis, which collec-tively, may reduce disease progression and improve brain activity. In addition, autologous adMSCs demonstrate low immunogenicity, which limits Graft Versus Host Disease (GVHD) during cell administration. Furthermore, our preclinical and clinical studies with adMSCs have shown that they are safe and effective at reducing inflammation and improving cognitive outcomes. A positive outcome would result in a paradigm shift in the treatment of AD that could potentially be a standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Has signed an informed consent form before any assessment is performed as part of the study.
2. Be male or female between 60 and 80 years old.
3. Subject has been or is in process of being clinically diagnosed with late pre-symptomatic or mild cognitive impairment (MCI) due to AD (prodromal AD).
4. Mini-Mental State Examination (MMSE) score of ≥ 22
5. Has an MRI to evaluate AD pathology (may use previous if within 6mo.)
6. Has APOE status to evaluate AD pathology (may use previous result)
7. Proficiency in English is required because cognitive tests are administered in English only.
8. Has evidence of brain amyloidosis via PET Scan or Aβ42/40 ratios in CSF.
9. Has evidence of peripheral inflammatory profile based on CRP (≥ 8 mg/L), IL-6 (≥ 3.1 pg/mL), TNF-α (10 pg/mL), or erythrocyte sedimentation rate (ESR) (≥20 mm/h) in blood assays.
10. Is in the opinion of the Investigator, in good general medical health based upon medical history, physical examination, laboratory tests, vital signs and EKG.

Exclusion Criteria:

1. Current medical or neurological condition that might impact cognition or performance on cognitive assessments. (e.g., traumatic brain injury (TBI), Parkinson's disease (PD), multiple sclerosis, etc.)
2. Inability or unwillingness of patient to undergo neuropsychological testing.
3. Advanced, severe, progressive or unstable disease that may interfere with the safety, tolerability and study assessments, or put the subject at special risk. (e.g., significant cardiac disease, severe renal impairment, severe hepatic impairment, autoimmune disease, etc.)
4. History of malignancy of any organ system within the past 60 months, that in the opinion of the investigator would impede evaluation or interpretation of subject safety or study results.
5. Females of childbearing potential must not be pregnant.
6. Inability or unwillingness to undergo PET Scans.
7. Inability or unwillingness to undergo MRI Scans.
8. Positive blood test for either HIV, Hepatitis B, Hepatitis C or Syphilis
9. Positive for TSPO SNP rs6971
10. Inability or unwillingness to undergo Lumbar Punctures.
11. Inability or unwillingness to undergo infusions.
12. Any condition, which in the opinion of the investigator, would put the subject at undue risk or would interfere with evaluation of the investigational product or interpretation of subject safety or study results.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in TSPO levels, measured by the PET scan, from baseline to midpoint and baseline to end of study | Baseline, midpoint (169 days from 1st infusion)
  Level of TSPO PET tracer will be measured for each PET scan. TSPO positivity, which is a marker for activated microglia, correlates with neuroinflammation
Inflammatory cytokines in CSF following adMSC therapy | Baseline, midpoint (169 days from 1st infusion)
  Inflammatory cytokine panel in CSF will be measured using commercially available immunosorbent assays to determine potential treatment effects. Aggregate values and percentages will be reported.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | Baseline - End of Study (337 days from 1st infusion)
  Safety endpoints will be monitored throughout the study and number of incidents reported at end of study. Aggregate values and percentages will be reported
Changes in neurofilament light chain (Nf-L) in CSF following adMSC therapy | Baseline, midpoint (169 days from 1st infusion)
  Levels of Nf-L in CSF will be measured using commercially available immunosorbent assays to determine potential treatment effects. Aggregate values and percentages will be reported.
Changes in Glial fibrillary acidic protein (GFAP) in CSF following adMSC therapy | Baseline, midpoint (169 days from 1st infusion)
  Levels of GFAP in CSF will be measured using commercially available immunosorbent assays to determine potential treatment effects. Aggregate values and percentages will be reported.
Changes in Total Tau/phosphor-Tau ratios in CSF following adMSC therapy | Baseline, midpoint (169 days from 1st infusion)
  Levels of Total Tau/phosphor-Tau ratios in CSF will be measured using commercially available immunosorbent assays to determine potential treatment effects. Aggregate values and percentages will be reported.
Changes in cerebral metabolism activity via FDG PET imaging from image baseline to midpoint | Baseline, midpoint (169 days from 1st infusion)
  Levels of [18F]FDG radiotracer will be measured for each PET scan. The uptake of [18F]FDG by the brain is a marker for cerebral metabolism activity
Changes in amyloid-β 42/40 ratio in CSF following adMSC therapy | Baseline, midpoint (169 days from 1st infusion)
  Levels of amyloid-β 42/40 ratio in CSF will be measured by LC/MS/MS assays. Aggregate values and percentages will be reported
Change in Mini-Mental Status Examination (MMSE) following adMSC therapy | Baseline, End of Study (337 days from 1st infusion)
  Cognition measured by MMSE. Scoring: 24-30 no cognitive impairment; 18-23 mild cognitive impairment; 0-17 severe cognitive impairment.
Change in Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) scores following adMSC therapy | Baseline, End of Study (337 days from 1st infusion)
  Cognitive decline measured by RBANS. Total Score subtest ranges: List Learning (0-40); Story Memory (0-24); Figure Copy (0-20); Line Orientation (0-20); Picture Naming (0-10); Semantic Fluency (4-40); Digit Span (0-16); Coding (0-89); List Recall (0-10); List Recognition (0-20); Story Recall (0-12); Figure Recall (0-20). Use Stimulus Booklet to convert Total Scores to Index Scores and Sum of Index Scores to Total Scale. Total Scores can range from 40 to 160. The RBANS scores are displayed as standard scores with means of 100 and a standard deviation of 15. Average/Mild Impairment (standard scores of 70 or above), Moderate Impairment (standard scores from 55 to 69), and Severe Impairment (standard scores <54).
Change in instrumental activities of daily living via Lawton IADL Scale scores following adMSC therapy | Baseline, End of Study (337 days from 1st infusion)
  The Lawton IADL scale contains eight items. Each ability measured by the scale relies on either cognitive or physical function, though all require some degree of both. The higher the score, the greater the person's abilities. Women are scored on all 8 areas of function, but, for men, the areas of food preparation, housekeeping, laundering are excluded. Clients are scored according to their highest level of functioning in that category. The final total score ranges from 0 (low function, dependent) to 8 (high function, independent) for women, and 0 through 5 for men. The final total score may be presented as a percentage of function. For example, a total score of 6 out of 8 would represent 75% function (75% independence, 25% dependence). Sequential scoring over time provides a measure of declining or
Measure immune pathway marker level changes in blood from screening/baseline to midpoint (D1-D169) and from screening/baseline to end of study (D1-D337) | Baseline, midpoint (169 days from 1st infusion), End of Study (337 days from 1st infusion)
  A commercially available immunological panel that tests markers associated with immunological pathways will be performed in blood at the end of study. Aggregate values and percentages will be reported.
Measure immune pathway marker level changes from screening/baseline to midpoint (D1-D169) in CSF | Baseline, midpoint (169 days from 1st infusion)
  A commercially available immunological panel that tests markers associated with immunological pathways will be performed in CSF at the end of study. Aggregate values and percentages will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Schulz, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston (UTHealth), Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No